CLINICAL TRIAL: NCT03471273
Title: Comparison of Endoscopic and Laparoscopic Resection for Small Gastric
Brief Title: Comparison of Endoscopic and Laparoscopic Resection for Small Gastric Gastrointestinal Stromal Tumor
Acronym: CELSGIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2016ZD013
Record Dates: First submitted 2018-01-19; First posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-01

CONDITIONS: Therapeutic Value of Endoscopic and Laparoscopic Resection for Small Gastric Gastrointestinal Stromal Tumor
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- endoscopic management (Other)
  Interventions: Procedure: endoscopic management, surgery and follow up
- follow up (Other)
  Interventions: Procedure: endoscopic management, surgery and follow up
- surgery (Other)
  Interventions: Procedure: endoscopic management, surgery and follow up

INTERVENTIONS:
Procedure: endoscopic management, surgery and follow up — endoscopic management, surgery and follow up

SUMMARY:
Comparison of Endoscopic and Laparoscopic Resection for Small Gastric Gastrointestinal Stromal Tumor

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old Chinese;
* Definite diagnosis or endoscopic ultrasonography, CT and other highly suspected Chinese patients with gastric stromal tumors;
* Patients voluntarily signed informed consent and have been orally informed of the specific trial plan.

Exclusion Criteria:

* Patients with gastric stromal tumors with distant metastasis who cannot be treated by laparoscopic surgery;
* Combined heart , cerebrovascular , liver , kidney , and hematopoietic system serious primary disease;
* gastric stromal tumors with severe digestive tract hemorrhage endanger the immediate surgical treatment of life;
* The investigator considers that it is not suitable for this test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
recur or not in 2 years after endoscopic surgical procedure or surgery | 2 years after endoscopic surgical procedure or surgery
  Participants will be followed up for 2 years after endoscopic surgical procedure or surgery by endoscope and/or endoscopic ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospistal, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided